CLINICAL TRIAL: NCT06576817
Title: Comparison of High-intensity Interval Circuit Training With Upper Extremity and Lower Extremity Training Versus Lower Extremity Training Alone in People With Parkinson Disease
Brief Title: High-intensity Interval Circuit Training in People With Parkinson Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-003
Record Dates: First submitted 2024-07-12; First posted 2024-08-29 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single center, two arm, pre-test post-test parallel design with up to 4 cohorts of class participants.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be told exercise stations may vary within-session and week to week but will not be informed that only one group has UE exercise interventions.
  Assessors are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower extremity and upper extremity exercise (Experimental): Exercises in the circuit (8 total) will focus on the lower extremity (4) and upper extremity (4)
  Interventions: Other: High intensity circuit exercise class - Lower and upper extremity
- Lower extremity exercise (Active Comparator): Exercises in the circuit (8 total) will focus on the lower extremity (4) alone.
  Interventions: Other: High intensity circuit exercise class - Lower extremity alone

INTERVENTIONS:
Other: High intensity circuit exercise class - Lower and upper extremity — Exercises performed at high intensity effort in the circuit (8 total) will focus on both the lower extremity (4) and upper extremity (4)
  Arms: Lower extremity and upper extremity exercise
Other: High intensity circuit exercise class - Lower extremity alone — All exercises performed at high intensity effort in the circuit (8 total) will focus on the lower extremity alone
  Arms: Lower extremity exercise

SUMMARY:
The goal of the study is to compare different types of high intensity circuit exercises over an 8-class training series in people with Parkinson disease. The main question it aims to answer is:

-Does including arm and hand exercises with leg exercises improve reaction time, balance, functional measures, gait speed and quality of life? This group will be compared to a group that only does leg exercises. Participants will be asked to participate in 8 high intensity circuit exercise classes.

DETAILED DESCRIPTION:
People with Parkinson disease will be recruited from the community and randomized into 2 equal groups: high intensity interval circuit training with lower extremity (LE) and lower and upper extremity (LEUE) training. The study will be composed of a baseline assessment, 8 group class sessions, and a post-intervention assessment. The baseline assessment will include demographics, disease and fall history and outcome measure collection. Group class sessions will include concurrent group warmup, followed by an 8-station circuit performed with high intensity intervals, and a cool-down. The circuit will include 4 stations performed by both the LE and LEUE groups and 4 stations specific to each intervention group, including 4 additional LE exercise stations for the LE group and 4 UE specific stations for the LEUE group. The stations that differ will not be adjacent to one another nor specifically indicated as different. The stations that differ will mirror similar aspects of function (ie, strength, reaction time, etc.) for the UE and LE stations. Participants will be told exercise stations may vary within-session and week to week but will not be informed that only one group has UE exercise interventions. After conclusion of the class series, post-intervention balance and stepping outcomes will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease
* Hoehn and Yahr level of 1 to 3
* ability to walk independently with or without an assistive device
* obtain medical clearance to participate in moderate or vigorous exercise.

Exclusion Criteria:

* diagnosis of any neurological disease other than PD (including but not limited to stroke, dementia, and multiple sclerosis; mild cognitive impairment is not excluded)
* bone instability (non-consolidated fractures, unstable spinal column, severe osteoporosis)
* muscle or ligament tears
* uncontrolled hypertension
* uncontrolled diabetes
* severe cardiovascular disease that impairs walking or exercise
* a major change in medication during the study training period (pre-test to post-test)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Trail making Test Parts A and B (timed, higher scores mean worse outcome) | 8-10 weeks
  Cognitive and fine motor skills
Activity-specific Balance Confidence Scale (0-100%, higher scores mean better outcome) | 8-10 weeks
  Balance confidence self-report
Timed Up and Go | 8-10 weeks
  Balance and function
10 meter Walk Test | 8-10 weeks
  Gait Speed
6 minute walk test | 8-10 weeks
  endurance
9-hole peg test (timed, higher scores mean worse outcome) | 8-10 weeks
  fine motor
Parkinson's Disease Questionnaire - Short Form (8) (Score 0-32, higher scores mean worse outcome) | 8-10 weeks
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany B Salido, DPT, PhD, Principal Investigator — Pacific Northwest University of Health Sciences
Locations (1):
- Pacific Northwest University of Health Sciences, Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: No